CLINICAL TRIAL: NCT02394613
Title: A Phase I, Storer Design, Open-label, Cross-sectional, Single Site Trial of ANX776 in Healthy Volunteers, Progressive Glaucoma/Glaucoma-suspect/Ocular Hypertensive Subjects and Non-arteritic Anterior Ischaemic Optic Neuropathy Subjects
Brief Title: A Phase I Clinical Trial of DARC
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University College, London (Other)
Collaborators: Wellcome Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 08/0351; 2014-002504-25 (EudraCT Number)
Record Dates: First submitted 2015-03-04; First posted 2015-03-20 (Estimated); Last update posted 2016-05-26 (Estimated); Status verified 2015-08

CONDITIONS: Glaucoma; Ocular Hypertension; Glaucoma, Suspect
Keywords: Glaucoma; DARC; Diagnosis
MeSH Terms: conditions — Glaucoma; Ocular Hypertension; Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- ANX776 (Experimental): Using and increasing dose storer design, GLAUCOMA and NORMAL patients will be randomly grouped to received the intervention (0.1 mg, 0.2 mg, 0.4 mg, 0.5 mg). 1 NAION patient will receive each dose once it has been proven safe in GLAUCOMA and NORMAL patients, as part of the secondary objective of this trial.
  Interventions: Drug: ANX776

INTERVENTIONS:
Drug: ANX776 — Single intravenous injection

SUMMARY:
Glaucoma is a major cause of irreversible blindness worldwide, caused by retinal nerve cell (RGC) death. This is currently identified only after significant vision loss has already occurred with an early event in, and a potential marker of, this process being RGC "apoptosis" (a form of cell death).

This study aims to investigate the tolerability and safety of ANX776, as part of the new Detection of Apoptosing Retinal Cells (DARC) technique. This has been developed by the laboratory of DARC IP holder and grant applicant: Prof. M. Francesca Cordeiro. A secondary aim is to initially establish the ability of DARC to identify RGC apoptosis in the diagnosis of glaucoma in healthy and progressive glaucoma/glaucoma-suspect/ocular hypertensive patients. As a positive control for this secondary aim of this study, patients with Non-arteritic Anterior Ischaemic Optic Neuropathy (NAION) will be recruited.

During the study, each patient will undergo several ophthalmological examinations, imaging of the back of the eye using established clinical devices, and blood sampling for studying the safety and toxicology profile of ANX776.

The understanding of the safety profile of ANX776 is crucial for the use of DARC in patients, and its application as a potentially powerful new clinical tool with which to identify patients with early glaucoma before their vision is lost. If successful, it opens the door to directly observing effects of glaucoma treatments, including the assessment of new, breakthrough therapies.

ELIGIBILITY:
Inclusion Criteria All patients

* ≥ 18 years
* Clear optical media in the studied eye
* No ocular or systemic disease (except glaucoma in the test group)
* Refractive error not higher than spherical equivalent of 6D; best corrected visual acuity ≥ 6/24 at qualification
* Proven ability to perform reliable visual field testing (HFA 640, central 24-2 program) to yield full thresholds, and have had good fundoscopy with assessment of the optic disc
* Willing and able to comply with the scheduled visits and assessments. Informed Consent Form personally (or by legal representative) signed and dated
* Women Not of Childbearing Potential (postmenopausal or permanently sterilised)
* Male participants agree to double barrier contraception from consent until 6 weeks after treatment discontinuation

GLAUCOMA patients

• Show progression in any measured parameter; have at least one eye with a diagnosis of glaucoma (abnormal optic disc, visual field defect or both); be diagnosed as a glaucoma suspect or ocular hypertensive (elevated Intraocular Pressure (IOP))

NORMAL subjects

* No evidence of any glaucomatous process (either optic disc, Retinal Nerve Fibre Layer (RNFL) of visual field abnormalities with normal IOPs)
* Must provide a GP letter confirming their medical history

GLAUCOMA & NORMAL patients • Have performed at least 3 Visual Field tests, Heidelberg Retinal Tomography (HRT), and Optical Coherence Tomography (OCT) before or during Visit-1

POSITIVE CONTROL patients

* Diagnosis of acute unilateral NAION in the first eye within 15 days of onset of symptoms
* Snellen test (or equivalent) Visual acuity below 6/12 in the affected eye
* Visual field defect and relative afferent pupillary defect (RAPD)
* Normal motility of the pupillary sphincter muscle
* Normal macula
* Completion of 1 Visual field test, OCT and HRT examination at Visit-1

Exclusion criteria All patients

* Terminal or mental illness, dementia, inability to comply with the study or follow-up procedures
* Presence of ocular or systemic uncontrolled disease (unless deemed not clinically significant by Chief Investigator and Sponsor), except glaucoma in the test group
* Central corneal thickness <450µm or >650µm
* History of current or severe, unstable or uncontrolled systemic disease (unless deemed not clinically significant by Chief Investigator and Sponsor)
* Body weight <40kg or >120kg
* Evidence of another chronic neurodegenerative condition
* Patients with active antiphospholipid syndrome or with diagnosis of circulating antiphospholipid antibodies
* History of clotting diseases (including Deep Vein Thromboses), subjects taking anticoagulants
* Diagnosis of thrombocytopenia, heart valve disease, and livedo reticularis
* Pregnancy or lactation
* Allergy to any study medication ingredient
* Inclusion in a clinical trial of an IMP within 12 weeks prior to study entry
* Ocular surgery within the past 3 months in the study eye
* History of retinal laser photocoagulation
* Media opacities or retinal pathology or amblyopia significantly limiting visual acuity, visual field test or retinal imaging
* Expected need for ocular surgery during the study
* Severe or acute or chronic medical or psychiatric condition or laboratory abnormality that, in the opinion of the Chief Investigator, makes the subject inappropriate for the study

GLAUCOMA patients

* Uncontrolled IOP >24 mmHg
* Angle closure/narrow glaucoma
* Mean deviation at Humphrey Visual Field (HVF) >12dB
* Unilateral glaucoma
* Secondary glaucoma

NORMAL subjects

* History of systemic vasculitis, collagenosis or ongoing treatment of cancer
* Active uveitis
* Evidence of previous retinal vascular disease

NORMAL & POSITIVE CONTROL subjects

• History or evidence of glaucoma (fundoscopy and Visual Field) or clinical suspicion of glaucoma on presentation or IOP ≥ 24 mmHg in either eye at any time

POSITIVE CONTROL patients

* Any other aetiology to explain optic nerve disease
* Evidence of giant cell arteritis (history, sedimentation rate)
* Evidence for other optic neuropathy (even fellow eye) or multiple sclerosis (history, clinical examination)
* History of other optic neuropathies
* History of NAION in the same eye
* Active/recurrent ocular inflammation that may prevent retinal imaging

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2015-05; Primary Completion 2015-11 (Actual); Study Completion 2016-08 (Estimated)

PRIMARY OUTCOMES:
Safety of ANX776 as defined by the number and nature of adverse events | 24 hours
  Serious and adverse medical events will be recorded

SECONDARY OUTCOMES:
DARC Count | 6 hours
  Confocal Laser-Scanning Ophthalmoscopy (cSLO) imaging will be used to ascertain the number of apoptosing retinal cells in each of the study populations.

CONTACTS AND LOCATIONS:
Overall Officials: Philip Bloom, MB ChB FRCS, Principal Investigator — Western Eye Hospital
Locations (1):
- Western Eye Hospital, Imperial College Healthcare NHS Trust,, London, United Kingdom